CLINICAL TRIAL: NCT05517811
Title: Use of Viscoelastic Assays Beyond Coagulation: Pre- and Post-operative TEG
Brief Title: Pre- and Post-operative TEG Indices in Patients With or Without Adenocarcinoma Undergoing Surgical Resection
Acronym: TEG
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-1844
Record Dates: First submitted 2022-08-04; First posted 2022-08-26 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Liver Cancer; Esophageal Cancer; Colorectal Cancer; Lung Adenocarcinoma; Control; Pancreas Cancer; Biliary Cancer
MeSH Terms: conditions — Liver Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms; Adenocarcinoma of Lung; Pancreatic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer: new diagnosis by the providing physician of hepatopancreaticobiliary, esophageal, colorectal or lung adenocarcinoma
  Interventions: Diagnostic Test: TEG indices
- Control: Patients undergoing major surgery
  Interventions: Diagnostic Test: TEG indices

INTERVENTIONS:
Diagnostic Test: TEG indices — Blood samples
  Other Names: Control

SUMMARY:
The investigators hypothesize that abnormalities in thromboelastography (TEG) parameters in patients with liver, pancreas, biliary, esophageal, colorectal, and lung adenocarcinoma can serve as biomarkers for oncologic disease burden, cancer recurrence and overall survival as well as thrombotic and hemorrhagic post-operative complications. The investigators further hypothesize that there is histologic pathology correlates to pre-operative TEG abnormalities, and that it identifies patients with virulent tumor biology.

DETAILED DESCRIPTION:
Aim 1: Evaluate the correlation between pre-operative TEG parameters and disease burden in patients with a new diagnosis of hepatopancreaticobiliary, esophageal, colorectal, and lung adenocarcinoma vs controls with no known malignancy.

Aim 2: Explore if pre- and post-operative TEG parameters vs routine clinical coagulation parameters (platelet count, prothrombin time [PT], partial thromboplastin time [PTT]) are predictive of pre- and post-operative thrombotic (deep vein thrombosis [DVT], pulmonary embolism [PE], stroke, myocardial infarct [MI]) and hemorrhagic complications.

Aim 3: Evaluate if correction of TEG parameters after surgery is predictive of curative resection and if the failure of TEG parameters to correct after surgery or chemoradiothearpy is predictive of cancer recurrence and overall survival.

Aim 4: Perform proteomic analyses on the tumor microenvironment of cancer tissue samples to investigate whether tumor histology and protein composition is associated with specific TEG derangements that have been previously correlated to poor outcomes, potentially identifying a specific subtype of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* new diagnosis by the providing physician of hepatopancreaticobiliary, esophageal, colorectal or lung adenocarcinoma will be eligible for enrollment in the study
* 18 Years and older

Exclusion Criteria:

* Under 18 years old
* prisoners
* those unable to provide informed consent
* pregnant women
* and those undergoing emergent or urgent operative intervention at the time of diagnosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are evaluated at the University of Colorado Cancer Center with a new diagnosis by the providing physician of hepatopancreaticobiliary, esophageal, colorectal or lung adenocarcinoma will be eligible for enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-06-26 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
TEG indices of coagulation | One Year
  R time (minutes ~ coagulation factors), angle (degrees ~ fibrinogen function), MA (mm ~ platelets function), and LY30 (%~ fibrinolysis) measured at baseline (initial presentation or time of diagnosis), after neoadjuvant chemotherapy (if applicable), pre-operatively (before the induction of general anesthesia), intra-operatively (after tumor removal), post-operative days 1, 3 and 5, and at routine follow up appointments at 2 weeks, 3 months, 6 months and 1 year after surgery.
Disease burden as measured by TNM staging | One year
  Disease burden as measured by TNM staging
Pre- operative thrombotic and hemorrhagic complications. | One Year
  Pre-operative thrombotic and hemorrhagic complications.
Recurrence free and overall survival. | One Year
  Recurrence free and overall survival.
Proteomic analysis of intro-operative sample tumor microenvironment | One Year
  Proteomic analysis of intro-operative sample tumor microenvironment
Post-operative thrombotic and hemorrhagic complications | One Year
  Post-operative thrombotic and hemorrhagic complications

SECONDARY OUTCOMES:
Tumor Type | One Year
  Benign, pre-malignant, malignant
Number of patients with pre-operative nodal | One Year
  Benign, pre-malignant, malignant
Number of patients withneuronal invasion | One year
  neuronal invasion
Number of patients with mass resectability | One year
  mass resectability
Number of patients withcomplete pathologic resection | one year
  complete pathologic resection
Number of patients withsurgical margins | One year
  surgical margins
blood transfusion requirements | One Year
  Number of patients withblood transfusion requirements
pre-operative distant metastasis | One year
  Number of patients withpre-operative distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gleisner, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided